CLINICAL TRIAL: NCT02844686
Title: Feasibility of Dynamic Cardiac SPECT With 99mTc-diethylenetriaminepenta-acetate (DTPA) for the Assessment of Myocardial Flow Reserve Using a Cadmium-Zinc-Telluride (CZT) Camera
Brief Title: Myocardial Flow Reserve and 99mTc-DTPA Cardiac Dynamic SPECT
Acronym: Flow-Heart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-004; 2016-000119-34 (EudraCT Number)
Record Dates: First submitted 2016-07-21; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial perfusion imaging; Single-Photon Emission Computer-Assisted Tomography
MeSH Terms: conditions — Coronary Artery Disease

ARMS (1):
- Cardiac Dynamic SPECT (Experimental)
  Interventions: Other: Cardiac SPECT

INTERVENTIONS:
Other: Cardiac SPECT — 3-D dynamic acquisition of cardiac SPECT at rest and after pharmacological stress

SUMMARY:
New CZT-based SPECT cameras are potentially capable of dynamic 3-D acquisition. Preliminary results suggested that dynamic acquisitions could allow the assessment of myocardial flow reserve using 99mTc-labelled perfusion tracers. The Flow-Heart study will assess the feasibility of myocardial flow reserve measurement by means of 99mTc-DTPA dynamic cardiac SPECT in 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patient clinically stable with known or suspected coronary disease
* Patient referred to Caen University Hospital for a myocardial perfusion SPECT
* Patient who accept to undergo subsequent additional cardiac dynamic SPECT using 99mTc-DTPA at rest and during pharmacological stress
* Informed consent dated and signed
* Affiliation to a social security system

Exclusion Criteria:

* Contraindication to dipyridamole (asthma, chronic obstructive pulmonary disease , pulmonary hypertension)
* History of poor tolerance of dipyridamole injection
* Cardiac arrhythmia (atrial fibrillation or frequent premature ventricular complex)
* Left bundle branch block, cardiac pacemaker, or implantable automatic defibrillator
* Recent history of myocardial infarction or unstable angina
* Pregnancy or lactating women
* Known obstructive renal or urinary disease
* Age under 18 years or guardianship
* Patient with an acute coronary syndrome or a coronary revascularization occurring between the conventional perfusion SPECT and the subsequent 99mTc-DTPA dynamic SPECT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of myocardial flow reserve assessment by dynamic cardiac SPECT using a CZT camera and 99mTc-DTPA | Within one month after a conventional myocardial perfusion SPECT

CONTACTS AND LOCATIONS:
Overall Officials: Alain Manrique, MD, PhD, Principal Investigator — University Hospital, Caen